CLINICAL TRIAL: NCT02839590
Title: The Effect of Glaucoma Surgery on Aqueous Dynamics in Patients With Glaucoma or Ocular Hypertension: An Observational Study
Brief Title: Aqueous Dynamics and Glaucoma Surgeries
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 163050; 15/LO/1809 (Other: Research Ethics Committee)
Record Dates: First submitted 2016-06-28; First posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Ocular hypertension; Aqueous dynamics
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Glaucoma Drainage Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- HiFu (ultrasound): Manufacturer Name Eyehope Principle intended use Surgical treatment of uncontrolled glaucoma and OHT The device is currently routinely used in the department for the treatment of uncontrolled glaucoma and OHT, and will be used in accordance with usual clinical practice. It is not anticipated that there will be any changes to the device or its usage during the course of the study.
  Interventions: Device: HiFU
- Baerveldt implant: Manufacturer Name Abbott Medical Optics Inc., Abbott Laboratories Inc., Abbott Park, Illinois, USA.
  Principle intended use Surgical treatment of uncontrolled glaucoma and OHT
  The device is currently routinely used in the department for the treatment of uncontrolled glaucoma and OHT, and will be used in accordance with usual clinical practice. It is not anticipated that there will be any changes to the device or its usage during the course of the study.
  Interventions: Device: Baerveldt implant
- Ahmed Implant: Manufacturer Name New World Medical, Inc., 10763 Edison Court, Rancho Cucamonga, CA 91730, USA.
  Principle intended use Surgical treatment of uncontrolled glaucoma and OHT
  The device is currently routinely used in the department for the treatment of uncontrolled glaucoma and OHT, and will be used in accordance with usual clinical practice. It is not anticipated that there will be any changes to the device or its usage during the course of the study.
  Interventions: Device: Ahmed implant
- STARflo: Manufacturer Name iSTAR Medical SA, Parc Créalys, Rue Phocas Lejeune, Bâtiment Regain 25/3, 5032 Isnes, Belgium.
  Principle intended use Surgical treatment of uncontrolled glaucoma and OHT
  The device is currently routinely used in the department for the treatment of uncontrolled glaucoma and OHT, and will be used in accordance with usual clinical practice. It is not anticipated that there will be any changes to the device or its usage during the course of the study.
  Interventions: Device: STARflo
- Hydrus Microstent implant: Manufacturer Name Ivantis, Inc., 38 Discovery, Suite 150, Irvine, CA 92618, USA.
  Principle intended use Surgical treatment of uncontrolled glaucoma and OHT
  The device is currently routinely used in the department for the treatment of uncontrolled glaucoma and OHT, and will be used in accordance with usual clinical practice. It is not anticipated that there will be any changes to the device or its usage during the course of the study.
  Interventions: Device: Hydrus Microstent implant
- iStent implant: Manufacturer Name Glaukos Corporation, 26051 Merit Circle, Suite 103, Laguna Hills, CA 92653, USA.
  Principle intended use Surgical treatment of uncontrolled glaucoma and OHT
  The device is currently routinely used in the department for the treatment of uncontrolled glaucoma and OHT, and will be used in accordance with usual clinical practice. It is not anticipated that there will be any changes to the device or its usage during the course of the study.
  Interventions: Device: iStent implant
- Kahook Dual Blade: Manufacturer: New World Medical. Inc. Single use, ophthalmic blade Utilizes ab interno approach through a clear cornea micro incision Dual blades positioned for precise parallel incisions of the trabecular meshwork with minimal residual leaflets Maintains natural physiologic outflow pathways
  Interventions: Device: Kahook Dual Blade

INTERVENTIONS:
Device: HiFU — Ciliary Ablation Treatment ( HiFu ultrasound treatment)
  Groups: HiFu (ultrasound)
Device: Baerveldt implant — External (sub-conjunctival) Drainage Surgery (Baerveldt implant)
  Groups: Baerveldt implant
Device: Ahmed implant — External (sub-conjunctival) Drainage Surgery (Ahmed Implant)
  Groups: Ahmed Implant
Device: STARflo — Suprachoroidal Shunt Surgery (STARflo)
  Groups: STARflo
Device: Hydrus Microstent implant — Trans-trabecular meshwork implants (Hydrus Microstent implant).
  Groups: Hydrus Microstent implant
Device: iStent implant — Trans-trabecular meshwork implants (iStent implant).
  Groups: iStent implant
Device: Kahook Dual Blade — It removes part of the trabecular meshwork
  Groups: Kahook Dual Blade

SUMMARY:
There are currently many surgical options for patients with glaucoma and ocular hypertension (OHT), including the Hydrus Microstent implant, HiFU (High intensity Focused ultrasound), STAR flo, Kahook Dual Blade, Diode laser, trabeculectomy and the Baerveldt implant, but little is known about how these different surgical techniques used to treat glaucoma affect the flow of fluid through and out of the eye (aqueous dynamics).

DETAILED DESCRIPTION:
Trial objectives

Main outcome measures: The following aqueous dynamics parameters will be measured: IOP, aqueous flow rate, trabecular outflow facility and uveoscleral outflow. These parameters will be measured pre-treatment (up to 2 months before glaucoma surgery) and repeated 3 months and 12 months post-surgery. Measures will be taken from the operated eye and the contra lateral non-operated eye which will be used as the control.

Trial design

This is a prospective observational study with the contra lateral untreated eye being used as control. Baseline measures will be conducted at a routine clinic visit up to 2 months before glaucoma surgery after 4 weeks of treatment washout.

Post-treatment follow-up measurements of the main outcomes will be conducted 3 months and 12 months after surgery, again, after 4 weeks wash out. A number of additional eye tests will also be performed to collect data for the study at the pre-operative appointment when the baseline measurements are taken and at the post-operative follow-up appointments 3 months and 12 months after the surgery. Other data will be collected from eye tests that are routinely performed pre-operatively and at the post-operative follow-up appointments 1 day, 1 week, 1 month, 3 months, 6 months, and 12 months after their surgery.

Study participants will be recruited from patients attending the Ophthalmology Department Outpatients Clinic at St Thomas' Hospital, London, United Kingdom who have a diagnosis of glaucoma or OHT (ocular hypertension) requiring glaucoma drainage surgery. One hundred patients with glaucoma or OHT and where a clinical decision has been made that they need glaucoma surgery will be included in the study such that 100 eyes undergoing surgery will be included together with the contra-lateral untreated eyes that will be used as controls for comparison with the treated eyes.

Data will be collected for the study at the following routine appointments that patients undergoing glaucoma surgery are asked to attend: a pre-operative appointment, surgery, and follow-up assessments 1 day, 1 week, 1 month, 3 months, 6 months, and 12 months after surgery. Baseline measurements will be taken up to 2 months before glaucoma surgery.

At the baseline assessment demographic information will be collected

Details of participants' relevant past medical history will be collected at the baseline pre-operative assessment and at 12 months post-surgery.

All tests will be performed on both eyes as the contra-lateral non-operated eye will be used as control.

Aqueous parameters

• Aqueous flow rate: Participants will be asked to self-administer 3 to 6 drops (depending on their age) of fluorescein sodium 2% topically into both eyes at 5 minute intervals on the night before the fluorophotometric scans. Fluorophotometry will be performed using a scanning ocular fluorophotometer from 9:00 am -12:00 midday. Four sets of triplicate scans will be collected at 1 hour intervals to determine the aqueous flow rate (Ft). The 3 scans are done in quick succession, taking approximately 2 seconds in total to complete the set. Following each set of scans, IOP will be measured using pneumatonometry. and rebound tonometry. IOP will be recorded as the mean of a total of 12 measurements per eye: 3 measurements every hour alternating between eyes.

Patients who have had previous cataract surgeries or iridotomy/iridectomy will be excluded from this aspect of the measurements as fluorophotometry is inaccurate in these eyes.

* Outflow facility: Tonographic outflow facility (C) measurement will be performed using an electronic Schiøtz tonographer (Model 720, Berkeley Bioengineering Inc, USA) between 9:00 am -12:00 midday. The facility of outflow will be measured from the rate of decay of IOP in the supine position during application of a recording Schiøtz tonometer over a period of 4 minutes with a standard 5.5 gram weight. The "R" values of the curve at every 30-second time point will be manually entered into the McLaren tonography computer program. The program fits a second-degree polynomial by least squares to the nine data points and determines the best-fit values for time 0 and time 4 minutes by extrapolation.
* Intraocular pressure (IOP): Pneumatonometry and rebound tonometry will be used to measure IOP for patients undergoing fluorophotometry. The IOP measurements will be recorded at 1 hour intervals between the hours of 9:00 am -12:00 midday following each set of fluorophotometric scans.
* Uveoscleral outflow: There are currently no reliable clinical methods of measuring uveoscleral outflow (Fu) and episcleral venous pressure (Pv). Fu will be therefore calculated using the Goldmann equation (see below) with an assumed episcleral venous pressure of 8-11 mmHg:

Ft = C(IOP - Pv) +Fu Where:

Ft = Measured aqueous flow rate Fu = Ft - C(IOP - Pv) Fu = Calculated uveoscleral outflow C = Tonographic outflow facility (value computed by the measurement device) IOP = Mean morning intraocular pressure as measured by pneumatonometry Pv = Episcleral venous pressure (8-11 mmHg, exact value calculated based on patient parameters)

Routine tests

At the pre-operative visit when baseline measurements are taken and at each routine post-operative follow-up visit (1 day, 1 week, 1 month, 3 months, 6 months, and 12 months after surgery) patients will undergo a clinical ophthalmological examination including the following tests and examinations:

* Visual acuity measurement (Snellen and ETDRS charts will be used. Best Corrected Distance Visual Acuity (BCVA) and Non Corrected Distance Visual Acuity (NCVA) will be measured using ETDRS (early treatment diabetic retinopathy study) charts. Best Corrected Near Visual Acuity (BCVA) will be measured using a standard near vision chart).
* Slit lamp examination
* Visual fields
* IOP (intraocular pressure) measurement (Goldmann applanation tonometry will be used to measure IOP, except when there is irregular corneal astigmatism or other corneal problems which may preclude accurate reading. The IOP measurement will be done after application of topical anesthetic (eye drop) with fluorescein)
* Gonioscopy
* Dilated fundoscopy
* Anterior chamber depth and axial length
* Central corneal thickness
* Refraction (routine at baseline only)

Description of the surgical interventions

There are potentially four types of operation that patients may have as part of their glaucoma care in the department:

* Trans-trabecular meshwork implants (Hydrus implant or iStent implant)
* Ciliary Ablation Treatment (Diode laser or HiFu ultrasound treatment)
* External (sub-conjunctival) Drainage Surgery (Trabeculectomy, Baerveldt implant or Ahmed Implant)
* Suprachoroidal Shunt Surgery (STARflo)

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 18 and 90 (inclusive).
* Able to understand the study and give informed consent.
* Willing, able and available to participate in all aspects of the study.
* Diagnosis of glaucoma or OHT which requires glaucoma surgery. (Defined as primary or secondary glaucoma; all types of secondary glaucoma may be included. Glaucoma will be diagnosed based on abnormal visual field testing and corresponding disc changes once seen by a glaucoma specialist.)
* Able to undergo accurate fluorophotometry and tonography.

Exclusion Criteria:

* Mental impairment conflicting with informed consent or follow-up.
* Allergy to fluorescein.
* Current use of any investigational drug or device or current participation in an interventional clinical trial.
* Patients who might not adequately understand written information given in English or verbal explanations in English will not be included as participants in the study must be able to understand English to complete some of the tests.
* Any inclusion criteria not met

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred patients with glaucoma or OHT and where a clinical decision has been made that they need glaucoma surgery will be included in the study such that 100 eyes undergoing surgery will be included together with the contralateral untreated eyes that will be used as controls for comparison with the treated eyes
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of Intraocular pressure at 12 months | baseline and 12 months
  It would be measured by Goldmann tonometer, iCare and pneumatonometer. The unit of measurement for all of these devices is the same. It is mmHg
Change from baseline of aqueous flow at 12 months | baseline and12 months
  This parameter is measured by fluorophotometry
Change from baseline of uveoscleral outflow at 12 months | baseline and 12 months
  It would be calculated by Goldmann's equation
Change from baseline of trabecular outflow facility at 12 months | baseline and 12 months
  It will be measured by Electronic Schiotz tonography

CONTACTS AND LOCATIONS:
Overall Officials: K Sheng Lim, MD, Principal Investigator — Guy's and St Thomas NHS Foundation Trust
Locations (1):
- St Thomas Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD)

REFERENCES:
- [Derived] Ho H, Daas A, Ho J, Alaghband P, Galvis EA, de Antonio Ramirez A, Grassi P, Lim R, Lim KS. Intraocular pressure changes following topical ocular hypotensive medications washout. Br J Ophthalmol. 2021 Feb;105(2):205-209. doi: 10.1136/bjophthalmol-2019-315778. Epub 2020 Apr 10. PMID 32277009